CLINICAL TRIAL: NCT02721082
Title: Changing the Default for Tobacco Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001774; R01HL131512 (NIH)
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Results first posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Tobacco Use Cessation
Keywords: tobacco treatment
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Nicotine Replacement Therapy; Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Opt Out (Experimental): Participants in this arm will be first enrolled to receive cessation treatment and will only not receive it by "opting out". Participant will receive a Opt Out treatment program. Participants will receive counseling and nicotine replacement therapy.
  Interventions: Behavioral: Opt Out Treatment Program; Drug: Nicotine Replacement Therapy
- Opt In (Active Comparator): Traditional approach to tobacco treatment program. Participants must first indicate they are ready to quit smoking by "opting in" to receive Opt In treatment program.
  Interventions: Behavioral: Opt In Treatment Program; Drug: Nicotine Replacement Therapy

INTERVENTIONS:
Behavioral: Opt Out Treatment Program — Tobacco Treatment (UKanQuit) staff will complete a treatment plan for all participants.
  Arms: Opt Out
Drug: Nicotine Replacement Therapy — Unless they Opt Out all participants will be provided with a 14 day supply of the nicotine patch and nicotine mini-lozenges or nicotine gum, depending on study related criteria.
  Other Names: Nicotine patch; Nicotine mini-lozenges; Nicotine gum
  Arms: Opt Out
Behavioral: Opt In Treatment Program — Tobacco Treatment (UKanQuit) staff will complete a treatment plan for participant's who are ready to quit smoking. For patient's not ready to quit, motivational counseling will be provided to participants based on principles of Motivational Interviewing.
  Arms: Opt In
Drug: Nicotine Replacement Therapy — Participants ready to quit will be provided with a 14 day supply of the nicotine patch and nicotine mini-lozenges or nicotine gum, depending on study related criteria.
  Other Names: Nicotine patch; Nicotine mini-lozenges; Nicotine gum
  Arms: Opt In

SUMMARY:
The purpose of this study is to determine the impact and efficacy of a new approach to smoking cessation treatment versus the traditional approach.

DETAILED DESCRIPTION:
In many health conditions, the default treatment approach is to first identify the health condition and then begin treatment. In this scenario, the physician discusses treatment options with the patient. The patient is free to decline treatment as they wish. If patients do nothing though, they will receive care.

For tobacco users, the default treatment is for them to "opt in" to receive smoking cessation assistance. The provider asks the smoker if they are ready to quit, and they offer medication and support only to those who respond back "yes". This limits the amount of smokers that receive treatment because only 1 in 3 smokers say they are ready to quit.

This study is looking at a novel approach to smoking cessation treatment. This study will compare the traditional, "standard of care" approach to opting in against a new approach where all smokers are provided with cessation medication and counseling unless they refuse it.

ELIGIBILITY:
Inclusion Criteria:

* Speak English or Spanish
* Have access to a telephone or mobile phone
* Not be currently pregnant or breast feeding
* Have no significant co-morbidity that precludes participation
* Current daily smoker
* Not in treatment for tobacco dependence
* Reside in Kansas or Missouri

Exclusion Criteria:

* Admission greater than 3 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimber Richter, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Richter KP, Catley D, Gajewski BJ, Faseru B, Shireman TI, Zhang C, Scheuermann TS, Mussulman LM, Nazir N, Hutcheson T, Shergina E, Ellerbeck EF. The Effects of Opt-out vs Opt-in Tobacco Treatment on Engagement, Cessation, and Costs: A Randomized Clinical Trial. JAMA Intern Med. 2023 Apr 1;183(4):331-339. doi: 10.1001/jamainternmed.2022.7170. PMID 36848129
- [Derived] Faseru B, Mussulman LM, Nazir N, Ellerbeck EF, Shergina E, Scheuermann TS, Gajewski BJ, Catley D, Richter KP. Use of pre-enrollment randomization and delayed consent to maximize participation in a clinical trial of opt-in versus opt-out tobacco treatment. Subst Abus. 2022;43(1):1035-1042. doi: 10.1080/08897077.2022.2060441. PMID 35435813
- [Derived] Faseru B, Ellerbeck EF, Catley D, Gajewski BJ, Scheuermann TS, Shireman TI, Mussulman LM, Nazir N, Bush T, Richter KP. Changing the default for tobacco-cessation treatment in an inpatient setting: study protocol of a randomized controlled trial. Trials. 2017 Aug 14;18(1):379. doi: 10.1186/s13063-017-2119-9. PMID 28806908

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Opt Out | Opt In
Started | 655 | 345
Completed | 469 | 270
Not Completed | 186 | 75

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opt Out | Opt In | Total
Number analyzed (Participants) | 469 | 270 | 739
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.21 (14.80) | 51.70 (14.56) | 51.39 (14.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226 | 123 | 349
  Male | 243 | 147 | 390
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 270 | 158 | 428
  Non-Hispanic Black | 83 | 49 | 132
  Non-Hispanic multiracial | 75 | 51 | 126
  Hispanic | 32 | 11 | 43
Region of Enrollment [Number; unit: participants]
  United States | 469 | 270 | 739

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point-prevalence Abstinence
Description: 7-day, self-reported and verified cigarette abstinence.
Time Frame: Month 1
Population: We calculated the Bayesian Posterior Probability (BPP) and Bayesian 95% Credible Intervals for all outcomes. ClinicalTrials.gov has no option to select these, so the labels for the credible intervals will appear as "confidence intervals"
Measure: Mean (95% Confidence Interval); unit: Percentage of participants quit at 1-mo
Arm/Group | Opt Out | Opt In
Number analyzed (Participants) | 469 | 270
Percentage of participants quit at 1-mo | 21.5 [17.9 to 25.4] | 15.8 [11.8 to 20.5]

2. Secondary Outcome: Treatment Engagement
Description: Percentages of participants who use cessation medications and participate in counseling post discharge
Time Frame: Month 1
Population: Accepted a post-discharge script for medication
Measure: Mean (95% Confidence Interval); unit: Percentage of participants w/script
Arm/Group | Opt Out | Opt In
Number analyzed (Participants) | 469 | 270
Percentage of participants w/script | 87.68 [84.50 to 90.54] | 37.84 [32.18 to 43.75]

3. Secondary Outcome: Default-theory Based Measures
Description: We will assess the impact of opt-out versus opt-in treatment on perceived treatment coercion using items adapted from the Admission Experience Survey (AES) short form.
Time Frame: Month 1
Population: BPP and credible intervals
Measure: Mean (95% Confidence Interval); unit: % felt they had control over quitting
Arm/Group | Opt Out | Opt In
Number analyzed (Participants) | 469 | 270
% felt they had control over quitting | 88.41 [85.19 to 91.28] | 86.64 [82.07 to 90.63]

4. Secondary Outcome: 7-day Point-prevalence Abstinence
Description: 7-day, self-reported and verified cigarette abstinence.
Time Frame: Month 6
Measure: Mean (95% Confidence Interval); unit: Percentage of participants quit at 6-mo
Arm/Group | Opt Out | Opt In
Number analyzed (Participants) | 469 | 270
Percentage of participants quit at 6-mo | 18.57 [15.0 to 22.4] | 17.90 [13.2 to 23.1]

5. Other Pre Specified Outcome: Cost-effectiveness
Description: Counselor time, wage estimates, pharmacotherapy costs, and abstinence rates will be combined to report the incremental cost-effective ratio (ICER). The ICER is the ratio of the difference in costs divided by the difference in effectiveness between the two study arms. ICER indicates the added cost per additional quitter, a metric that will allow comparisons to other smoking cessation economic studies.
Time Frame: Month 6
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collect for 6 months following randomization
Description: Definitions do not differ from those of clinicaltrials.gov
Arm/Group | Opt Out | Opt In
All-Cause Mortality (participants affected / at risk) | 27/655 | 19/345
Serious Adverse Events (participants affected / at risk) | 191/655 | 89/345
Other Adverse Events (participants affected / at risk) | 0/655 | 0/345
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opt Out (N=655) | Opt In (N=345)
Death, Hospitalization, or Life threatening illness (General disorders) | 191 (191) | 89 (89) — Most adverse events were repeat hospitalizations, which is common in a population recruited during hospital admission

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT02721082/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT02721082/SAP_001.pdf